CLINICAL TRIAL: NCT02260232
Title: Worksite Exercise Intervention Effects on Cardiovascular Disease Risk Factors and Physical Activity Levels Among Healthy Employees
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Europea de Madrid (Other)
Responsible Party: Principal Investigator, Oscar Garcia Lopez, Professor, Universidad Europea de Madrid
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: UEM_ASISA_1
Record Dates: First submitted 2014-10-06; First posted 2014-10-09 (Estimated); Last update posted 2014-10-09 (Estimated); Status verified 2014-10

CONDITIONS: Exercise Therapy
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- exercise intervention (Experimental): Components of the program included supervised moderate to high intensity cardiorespiratory exercise, resistance training, and flexibility.
  Interventions: Other: exercise training
- control (No Intervention)

INTERVENTIONS:
Other: exercise training
  Arms: exercise intervention

SUMMARY:
Objective: To investigate the effects of a one-year worksite individual exercise intervention on lifestyle-related modifiable health risks, physical capacity and work performance.

Methods: Two hundred ninety-five employees volunteered to participate (n=191 women, n=104 men), aged 38 ± 8 years and body mass index (BMI), 24.71 ± 3.79. Measures of physical activity levels were assessed by the long self-administrated version of the International Physical Activity Questionnaire-Long Form (IPAQ-L), and all subjects performed a maximal cardiopulmonary treadmill graded exercise test. Blood samples and anthropometry measures were collected from participants at baseline survey, at 6 months and 1-year after. Components of the program included supervised moderate to high intensity cardiorespiratory exercise, resistance training, and flexibility.

ELIGIBILITY:
Inclusion Criteria:

Working in ASISA company, middle-age (20-60)

Exclusion Criteria:

No medical condition contraindicating exercise participation

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 295 (Actual)
Dates: Start 2010-06; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
International Physical Activity Questionnaire-Long Form (IPAQ-L) | 1 week
Graded cardiorespiratory fitness exercise test | 1 week